CLINICAL TRIAL: NCT06199479
Title: Radiologic Pathologic Correlation of Imaging to Distinguish True Progression From Pseudoprogression in Brain Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0671; NCI-2023-11127 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Brain Malignancies; Pseudoprogression
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): The tests and procedures done as part of your standard-of-care biopsy preparation, participants will also have advanced MRI and CT scans performed no later than 2 weeks before the biopsy. Typically, these scans are done within 1 or 2 days before surgery to provide the most accurate images to the surgeon.
  Interventions: Procedure: MRI Scan; Procedure: CT Scan; Procedure: Biopsy

INTERVENTIONS:
Procedure: MRI Scan — Performed by MRI Scan
Procedure: CT Scan — Performed by CT Scan
Procedure: Biopsy — Standard of Care Biopsy

SUMMARY:
To learn if advanced imaging methods can tell apart true progression (the disease has actually gotten worse) from pseudoprogression (the disease appears to have gotten worse, but it actually has not).

DETAILED DESCRIPTION:
Primary Objectives To determine if advanced imaging findings can correlate with tissue changes in order to distinguish true progression from pseudoprogression. We will recruit participants with new suspicious enhancement developing during treatment for glioma, and systematically perform: a) high quality routine MR imaging (including routine, diffusion, permeability, perfusion and spectroscopy imaging as part of our regular ABTI protocol) and compare this imaging to b) pathology obtained by means of stereotactic biopsy. Pathology will serve as the gold standard to determine which imaging strategies are most successful in distinguishing between true Tumor recurrence and Pseudoprogression for each lesion.

Secondary Objectives

1. To assess the feasibility of Contrast Clearance MR (delayed T1 enhanced MR) subtraction maps in distinguishing Pseudoprogression from true progression.
2. To gather observational data for Dual Energy CT imaging and delayed contrast clearance with Dual Energy CT in the assessment of glioma.
3. To correlate quantitative imaging biomarkers (derived from MR imaging data) along the biopsy tract with histological and clinical biomarkers. This exploratory data could generate novel comparisons to determine those imaging biomarkers that are most effective at predicting (a) cellular density and, (b) the types and relative numbers of cells present in the brain.
4. To observe clinical outcomes such as progression free survival and overall survival in the trial population and relate these to imaging findings.

ELIGIBILITY:
Inclusion Criteria:

1. Participants is >18 years old. The pediatric population has a different disease profile from adult glioma participants. To reduce heterogeneity in the patient population we will not consider participants younger than 18 for this study.
2. The participants agrees to participate in the clinical study and to complete all required visits and evaluations.
3. Participants has undergone prior treatment for a brain tumor and has a new suspicious imaging finding requiring diagnostic workup and is being considered for biopsy.
4. Participants agrees to undergo, prior to the procedure, the needed imaging evaluation (within 14 days and preferably with 3 days of the planned procedure).

Exclusion Criteria:

1. Renal failure as evidenced by a GFR of less than 30 mL/min/1.73m2 for gadolinium based imaging. In the absence of eGFR lab result, participants is not excluded in the absence of remarkable pathological renal history, as confirmed by and in the discretion of the PI.
2. For iodinated contrast agent we will use the more strict cut-off of 45 mL/min/1.73m2 ((Davenport, Perazella et al. 2020), Consensus statement from the ACR and the National Kidney Foundation). The different threshold reflects the different risk profiles of these agents. Participants with GFR in the range 30-45 can receive a Non-Contrast DECT (CT contrast withheld).
3. Pacemakers, electronic stimulation, metallic foreign bodies and devices and/or other conditions that are not MR safe, which include but are not limited to:

   * electronically, magnetically, and mechanically activated implants
   * ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators and cardiac pacemakers
   * metallic splinters in the eye
   * ferromagnetic hemostatic clips in the central nervous system (CNS) or body
   * cochlear implants
   * other pacemakers, e.g., for the carotid sinus
   * insulin pumps and nerve stimulators
   * non-MR safe lead wires
   * prosthetic heart valves (if dehiscence is suspected)
   * non-ferromagnetic stapedial implants
   * pregnancy
   * claustrophobia that does not readily respond to oral medication.

   Nonetheless, if patients have an electronic device for which manufacturer's guidelines exist to permit safe MR scanning (such as the Cardiology supervised pacemaker scanning program), such a patient would still be eligible to participate in the trial. Such patients will be scanned as per manufacturers recommendations.
4. Allergy to relevant imaging contrast agents, includes allergies to iodine or gadolinium-based contrast agents (if one class of agents is contra-indicated, then imaging with the other can still proceed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Dawid Schellingerhout, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org